CLINICAL TRIAL: NCT02435082
Title: Vascular Assessment of Regulation Index Arrays Registry
Acronym: VARIA
Status: Completed | Type: Observational
Sponsor: NeuroChaos Solutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Varia-REG 1.0
Record Dates: First submitted 2015-04-20; First posted 2015-05-06 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Concussion
Keywords: Concussion; Vascular Assessment; Vascular Regulation; mild Traumatic Brain Injury, mTBI; Traumatic Brain Injury, TBI; Cerebrovascular Regulation; Cerebral Blood Flow; Cerebral Blood Flow Velocity, CBFV; Cerebral Blood Flow Velocity Variability; Cerebrovascular Assessment
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Concussion with TCD: Any patient (adolescent/adult) receiving a Transcranial Doppler (TCD) for a head injury, suspected concussion, or suspected mild traumatic brain injury (sports related or not).

SUMMARY:
The objective of this patient registry is to collect and analyze physiological data associated with baseline and brain injury identified in standard clinical practice (Normal Values, Recovery Curves, Correlation between Symptoms and Other Tests, NCI Index), and to assess health economics.

DETAILED DESCRIPTION:
The key aims of the VARIA Registry are to determine the real-life testing patterns and clinical outcomes of newly diagnosed patients with brain injury.

In accordance with the primary objective, the study will collect and analyze physiological data associated with brain injury identified in normal clinical practice with specific reference to:

* Patient demographics, symptoms, NCI Index, and other test results,
* Baseline ranges by demographic group,
* Post-injury patients presenting without a baseline test to be assessed in the context of the norms for similar patients,
* Recovery curves by demographic,
* Health Economics.

This registry will be a prospective observational study to collect data to describe the real-life testing patterns and clinical outcomes of newly diagnosed patients with brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Any patient receiving a Transcranial Doppler for a brain injury
* Adolescents and Adults
* Written informed consent obtained by the clinician (may not be required for retrospective cases)

Exclusion Criteria:

* Alcohol/substance abuse within the past 6 months, patient reported
* Serious mental illness that might preclude subject's ability to comply with treatment

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients contacting a clinic to schedule an appointment for evaluation of the brain (pre or post injury) will be informed about the registry and will be given the option to participate.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Neurovascular Complexity Index (NCI) measured by Varia-NCI | Baseline
  Patient Neurovascular Complexity Index (NCI) will be measured

SECONDARY OUTCOMES:
Neurovascular Complexity Index (NCI) measured by Varia-NCI | Every 4-7 days post injury; up to 6 months after injury resolution
  Patient Neurovascular Complexity Index (NCI) will be measured.
Cognition measured by clinical praxis | Every 4-7 days post injury; up to 6 months after injury resolution
  Patient cognitive status will be measured
Physiology measured by clinical praxis | Every 4-7 days post injury; up to 6 months after injury resolution
  Patient physiological status will be assessed
Cognition measured by clinical praxis | Baseline
  Patient cognitive status will be measured
Physiology measured by clinical praxis | Baseline
  Patient physiological status will be assessed

OTHER OUTCOMES:
Health Economic Outcomes measured by clinical praxis | Every 4-7 days post injury; up to 6 months after injury resolution
  Health economic parameters and consumption of resources will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Vladislav Bukhman, PhD, Study Chair — NeuroChaos Solutions
Locations (1):
- SportsSafe, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No